CLINICAL TRIAL: NCT04573179
Title: Effectiveness of 68Ga-PSMA PET/MRI for Improving the Detection of Clinical Significant Prostate Cancer in Lesions With Prostate Imaging Reporting and Data System Score 3
Brief Title: Effectiveness of 68Ga-PSMA PET/MRI for Improving the Detection of csPCa in Lesions With PI-RADS Score 3
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Principal Investigator, Hongqian Guo, Executive officer of Department of Urology, Drum Tower Hospital, Medical School of Nanjing University, Institute of Urology, Nanjing University, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Other Study IDs: AF/SQ-05/30
Record Dates: First submitted 2020-09-28; First posted 2020-10-05 (Actual); Last update posted 2020-10-05 (Actual); Status verified 2020-09

CONDITIONS: Prostatic Neoplasms
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study was to explore the effectiveness of 68Ga-PSMA PET/MRI for improving the detection of csPCa in lesions with PI-RADS score 3. This study is a prospective, observational study, single-center research. After recruiting patients who are suspected prostate cancer with a mpMRI PI-RADS version2 score of 3 and willing to perform prostate biopsy to identify the diagnosis, 68Ga-PSMA PET/MRI will be performed. Lesions will be reaccessed based on PET/MRI findings and compared with the pathological results.

ELIGIBILITY:
Inclusion Criteria:

* males over 18 years old suspected for prostate cancer
* serum PSA between 4ng/ml and 20ng/ml in recent two months
* mpMRI PI-RADS version2 scores 3 in recent two months
* willing to undertake prostate biopsy
* no evidence of non-cancerous factors interfere PSA level, such as catheter insertion, bladder stones, urinary tract infections or drug (e.g. finasteride)
* ECOG 0-1

Exclusion Criteria:

* history of prostate biopsy or other operations
* history of prostate cancer associated treatment
* contraindications for MRI or PET examination (e.g. claustrophobia, pacemakers, hip metal implants, hyperglycemia, glomerular filtration rate less than 50 ml/min)
* not suitable for prostate biopsy (e.g. coagulation dysfunction, skin infection at perineal puncture site)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: community residents
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-03-01 (Estimated); Study Completion 2021-07-01 (Estimated)

PRIMARY OUTCOMES:
detection rate | one year
  detection rate of csPCa

SECONDARY OUTCOMES:
detection rate | one year
  detection rate of non-csPCa

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Urology, Drum Tower Hospital, Medical School of Nanjing University, Institute of Urology, Nanjing University, Nanjing, Jiangsu, China